CLINICAL TRIAL: NCT03207269
Title: A High-protein Bedtime Snack to Control Morning Blood Glucose
Brief Title: Impact of Bedtime Snacks on Glucose Control in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H17-01055
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High protein no carbohydrate (Experimental): Dietary. Two eggs will be consumed 30 minutes prior to bedtime. Energy content of dinner will be reduced to account for the calories in the bedtime snack.
  Interventions: Other: Dietary
- High protein carbohydrate containing (Active Comparator): Dietary. A low-fat yogurt will be consumed 30 minutes prior to bedtime. Protein will be matched to the high protein bedtime snack condition. Energy content of dinner will be reduced to account for the calories in the bedtime snack.
  Interventions: Other: Dietary
- Control no snack (No Intervention): No snack will be consumed prior to bed.

INTERVENTIONS:
Other: Dietary — Diet will be manipulated by providing different bedtime snacks within an otherwise isocaloric diet.
  Arms: High protein carbohydrate containing; High protein no carbohydrate

SUMMARY:
Approximately 3 million Canadians have type 2 diabetes, a condition where the blood sugar levels are too high, uncontrolled blood sugars lead to cardiovascular disease and other complications. Patients with type 2 diabetes are often advised to consume a snack before bed in order to help control morning blood sugar levels. However, scientific evidence for this dietary approach is limited and there is no data to help elucidate what the ideal bedtime snack is. We hypothesize that a high protein, high fat snack with very little carbohydrate, will be an effective bedtime snack for lowering morning glucose without spiking glucose levels in the night. In this study we will determine if a bedtime snack that is high in protein and fat but low in carbohydrate can help improve morning glucose control in people with type 2 diabetes. This information will provide scientific evidence for the potential health benefits of strategically-timed high protein, high fat snack consumption in people with type 2 diabetes.

DETAILED DESCRIPTION:
Fifteen patients with physician diagnosed type 2 diabetes (HbA1c 6.5-9%), between the ages of 30-80 years, and not on exogenous insulin therapy, will complete three, 3-day intervention periods (proof-of-concept randomized trial). Participants will consume a standardized diet for three days with either i) two hard-boiled eggs, ii) fruit yogurt; or iii) control no-bedtime snack, thirty minutes prior to bedtime. Fasting blood samples will be obtained on Day 4 in the morning after following each 3-day dietary intervention. Blood glucose will be monitored continuously across the intervention period using continuous glucose monitoring (CGM). CGM allows for the moment-to-moment changes in blood glucose to be examined for several days, allowing the unique opportunity to examine the glucose responses at different points of the day, including fasting hyperglycemia in the morning, nocturnal glucose, and postprandial glucose in response to meals. To our knowledge, CGM technology has never been used in a bedtime snacking study in type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Type 2 Diabetes
* HbA1c between 6.5 - 9.0%
* No dietary restraints (lactose intolerance, dislike eggs, celiac disease)

Exclusion Criteria:

* Heart attack or stroke within last year
* Exogenous insulin

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma glucose | Day 4
  Fasting Plasma glucose

SECONDARY OUTCOMES:
24 h mean blood glucose | Average of three days during each intervention
  continuous blood glucose monitoring
postprandial glucose | Average of three days during each intervention
  breakfast AUC
Fasting insulin | Average of three days during each intervention
  Fasting plasma insulin
Fasting homeostasis model assessment of insulin resistance (HOMA-IR) | Day 4
  Calculated by fasting plasma glucose and insulin
Overnight blood glucose | Average of three days during each intervention
  Glucose assessed during sleep by continuous glucose monitoring
Fasting continuous glucose monitoring glucose | Average of the three days during each intervention
  15-minute average glucose assessed by CGM in the fasted state upon awakening

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbie E, Francois ME, Chang CR, Barry JC, Little JP. A low-carbohydrate protein-rich bedtime snack to control fasting and nocturnal glucose in type 2 diabetes: A randomized trial. Clin Nutr. 2020 Dec;39(12):3601-3606. doi: 10.1016/j.clnu.2020.03.008. Epub 2020 Mar 13. PMID 32204977